CLINICAL TRIAL: NCT00287326
Title: Comparison of Epidural Bupivacaine-Clonidine With Intravenous Morphine Versus Intravenous Morphine Alone for Post-Operative Pain Relief in Pediatric Patients Undergoing Lower Extremity or Pelvic Osteotomy.
Brief Title: Comparison of Low-dose Epidural With Intravenous Narcotic Versus Intravenous Narcotic Alone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated by PI
Sponsor: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-Anes-231
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: Epidural; Bupivacaine; Clonidine
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Clonidine; Morphine

INTERVENTIONS:
Drug: Bupivacaine, Clonidine, Morphine

SUMMARY:
The purpose of the study is to determine if a low-dose epidural drug mixture without narcotic will result in lower parenteral narcotic usage, and improved side-effect profile for post-operative pain in the pediatric population undergoing lower extremity or pelvic osteotomy.

DETAILED DESCRIPTION:
Post-operative pain in patients undergoing osteotomy can be severe. Current methods of treatment involve parenteral narcotics and regional anesthesia. Several studies have looked at the efficacy of regional anesthesia with various combinations of local anesthetic and additives in different populations. However, to our knowledge there have been none that directly compare bupivacaine/clonidine epidural with supplemental narcotics to parenteral narcotics alone. Many studies substantiate the efficacy of bupivacaine and clonidine as effective drugs for epidural analgesia (1,2,3). Parenteral narcotic alone is associated with the possibility of significant side effects, overdose, and inadequate analgesia. Epidural analgesia has been shown to reduce postoperative pain scores more than parenteral narcotics (4). We believe that this study is important since the protocol allows additional parenteral narcotic in the epidural group if needed, and also allows for narcotic dosing prior to discontinuation of the epidural to compensate for rebound pain. Further, the prolongation of pain control shown with epidural clonidine may be beneficial during the transition (5,6).

ELIGIBILITY:
Inclusion Criteria:

* Age 4-16
* English speaking
* Elective lower extremity osteotomy
* Expected length of stay greater than 24 hours

Exclusion Criteria:

* History of previous spine surgery
* Current infection overlying catheter insertion site
* Coagulopathy

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
24 hour recording of pain, sedation, narcotic usage, and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Stella, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States